CLINICAL TRIAL: NCT01818206
Title: Bacteriophages Effects on Pseudomonas Aeruginosa Presents in Sputum of Cystic Fibrosis (CF) Patients
Brief Title: Bacteriophage Effects on Pseudomonas Aeruginosa
Acronym: MUCOPHAGES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UF 8750
Record Dates: First submitted 2013-03-21; First posted 2013-03-26 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Bacteriophages; Pseudomonas aeruginosa; Sputum
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cystic fibrosis (CF) patients (Experimental): Cystic fibrosis patients whom induced sputum is collected in order to evaluate the efficacy of a cocktail of 10 bacteriophages.
  Interventions: Other: Collection of induced sputum in order to evaluate the efficacy of a cocktail of 10 bacteriophages.

INTERVENTIONS:
Other: Collection of induced sputum in order to evaluate the efficacy of a cocktail of 10 bacteriophages. — Collection of induced sputum on cystic fibrosis patients in order to evaluate the efficacy of a cocktail of 10 bacteriophages.

SUMMARY:
Pulmonary phage therapy to treat bacterial infections of the respiratory tract have been investigated in animals. The aim of the present study is to evaluate the efficacy of bacteriophages in infecting Pseudomonas aeruginosa (PA) strains present in sputum samples. A cocktail of 10 bacteriophages will be applied on 60 sputum samples obtained from cystic fibrosis (CF) patients during 6 hours.We will determine the bacteria and bacteriophages strains in sputum samples collected. Then the sensitivity of individual colony will be tested.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Affiliated or benefit from a disease insurance regimen
* Men and women
* Aged from at least 6 years old
* Confirmed Diagnosis of cystic fibrosis based on presence of 2 mutations of CFTR gene and/or 2 positive tests of sweat chloride and/or 2 measures of pathologic difference of nasal potential associated to cystic fibrosis clinical signs.
* Patients able to produce sputum
* Pseudomonas aeruginosa Chronic infected patients

Exclusion Criteria:

* Simultaneous participation to another project on anti-infection, anti-inflammatory or modificating agents
* Subjet in exclusion period
* Law protected patient
* Realisation of sputum production is contra-indicated

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Pseudomonas aeruginosa (PA) strains counts after 6 hours in presence of bacteriophage | after 6 hours in presence of bacteriophage

SECONDARY OUTCOMES:
Pseudomonas aeruginosa (PA) strains counts after 24 hours in presence of bacteriophage | after 24 hours in presence of bacteriophage
Bacteriophage counts after 6 hours incubation within sputum samples | after 6 hours incubation within sputum samples
Sensitivity of individual Pseudomonas aeruginosa (PA) colonies to bacteriophages | Sensitivity of individual PA colonies to bacteriophages

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël RC CHIRON, RC, Principal Investigator — CHU de Montpellier - Hôpital Arnaud de Villeneuve
Locations (1):
- CHU de Montpellier - Hôpital Arnaud de Villeneuve CRCM, Montpellier, Languedoc Roussillon, France